CLINICAL TRIAL: NCT04097600
Title: A Comparative Bioavailability Trial of Steady State Semaglutide Exposure With the Current Formulation (Semaglutide) and a New Formulation (Semaglutide D) of Oral Semaglutide in Healthy Subjects
Brief Title: A Research Study Comparing Active Drug in the Blood in Healthy Participants Following Dosing of the Current and a New Formulation (D) Semaglutide Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4486; U1111-1226-6257 (Other: World Health Organization (WHO)); 2019-000279-17 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Current form 3 mg in treatment period 1, followed by current form 7 mg in treatment period 2, followed by new form 11.2 mg in treatment period 3
  Interventions: Drug: Oral semaglutide
- Sequence 2 (Experimental): Current form 3 mg in treatment period 1, followed by new form 5.6 mg in treatment period 2, followed by current form 14 mg in treatment period 3
  Interventions: Drug: Oral semaglutide
- Sequence 3 (Experimental): New form 2.4 mg in treatment period 1, followed by current form 7 mg in treatment period 2, followed by current form 14 mg in treatment period 3
  Interventions: Drug: Oral semaglutide
- Sequence 4 (Experimental): New form 2.4 mg in treatment period 1, followed by new form 5.6 mg in treatment period 2, followed by current form 14 mg in treatment period 3
  Interventions: Drug: Oral semaglutide
- Sequence 5 (Experimental): New form 2.4 mg in treatment period 1, followed by current form 7 mg in treatment period 2, followed by new form 11.2 mg in treatment period 3
  Interventions: Drug: Oral semaglutide
- Sequence 6 (Experimental): Current form 3 mg in treatment period 1, followed by new form 5.6 mg in treatment period 2, followed by new form 11.2 mg in treatment period 3
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Oral semaglutide current formulation and oral semaglutide new formulation, each in 3 different strengths, administered once daily during 6 treatment periods, each lasting 12 weeks

SUMMARY:
In this study two different tablets for oral use of a known investigational medicinal product, called semaglutide, will be tested. One is the current formulation and the other one is a new formulation of semaglutide. Both will be administered as a tablet and are for the treatment of diabetes. Currently, semaglutide is only prescribed as injections for the treatment of diabetes in some countries. The aim of this study is to find out if the dosage strength of the current formulation of semaglutide can be reduced in the new tablet formulation. For this purpose, it will be measured how much semaglutide is taken up in the body from the two (2) different tablet formulations each with three (3) different dosage strengths. The tablet version of the study medicine is a new medicine that cannot yet be prescribed. Participants will either get semaglutide in the current tablet formulation previously tested in many large studies, or get the tablet that contains semaglutide in a new formulation - which treatment is decided by chance. Participants will get one tablet per day over 4 weeks in each of the 3 treatment periods (i.e. treatment in a total of 12 weeks). The tablets should be taken in the morning together with half a glass of water (120 mL), after an overnight fast of at least 6 hours (no food or drinks). Furthermore, water is not allowed from 2 hours before dosing. After dosing participants must wait 30 minutes before they may eat or drink. At home, participants must take their breakfast 30-45 minutes after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 kg/m^2 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Glycated haemoglobin (HbA1c) equal to or above 6.5 % (48 mmol/mol) at screening.
* Use of tobacco and nicotine products, defined as any of the below:
* Smoking more than 5 cigarettes or the equivalent per day
* Not willing to refrain from smoking and use of nicotine substitute products during the in-house period(s)
* History (as declared by the subject) of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by the subject).
* History (as declared by the subject) or presence of pancreatitis (acute or chronic).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 274 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,sema,SS; area under the semaglutide plasma concentration-time curve during a dosing interval at steady state | From 0 to 24 hours after the last dosing of oral semaglutide low, medium and high dose on days 28, 56 and 84, respectively
  nmol*h/L

SECONDARY OUTCOMES:
Cmax,sema,SS; maximum semaglutide plasma concentration at steady state | From 0 to 24 hours after the last dosing of oral semaglutide low, medium and high dose on days 28, 56 and 84, respectively
  nmol/L
tmax,sema,SS; time to maximum semaglutide plasma contraction at steady state | From 0 to 24 hours after the last dosing of oral semaglutide low, medium and high dose on days 28, 56 and 84, respectively
  h
t½,sema,SS; terminal half-life of semaglutide at steady state | Determined by concentrations measured between day 84 and follow-up at day 119 of semaglutide at steady state
  h

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com